CLINICAL TRIAL: NCT02614040
Title: Saline Against Lactated Ringers or Plasmalyte in the Emergency Department (SaLt-ED)
Brief Title: Saline Against Lactated Ringers or Plasmalyte in the Emergency Department
Acronym: SaLt-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Wesley Self, Associate Professor of Emergency Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151769
Record Dates: First submitted 2015-11-18; First posted 2015-11-25 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Critical Illness; Acute Kidney Injury
Keywords: crystalloid; acute kidney injury
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury | interventions — Saline Solution; Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9% Saline (Active Comparator): Patients in a month randomized to physiologically-balanced isotonic fluid will receive 0.9% Saline whenever isotonic intravenous fluid administration is ordered by the treating provider.
  Interventions: Other: 0.9% Saline
- Physiologically-balanced (Active Comparator): Patients in a month randomized to physiologically-balanced isotonic fluid will receive physiologically-balanced isotonic crystalloid (Plasma-Lyte© A or Lactated Ringer's) whenever isotonic intravenous fluid administration is ordered by the treating provider.
  Interventions: Other: Physiologically-balanced isotonic crystalloid

INTERVENTIONS:
Other: 0.9% Saline — 0.9% Saline will be used whenever an isotonic crystalloid is ordered
  Other Names: Normal saline; 0.9% sodium chloride
  Arms: 0.9% Saline
Other: Physiologically-balanced isotonic crystalloid — Lactated Ringers or Plasma-Lyte© A will be used whenever an isotonic crystalloid is ordered
  Other Names: Lactated Ringers; Ringer's Lactate; Plasma-Lyte© A
  Arms: Physiologically-balanced

SUMMARY:
This study will be a cluster-randomized, single-center trial comparing 0.9% saline (normal saline) vs physiologically-balanced crystalloid fluids (Lactated Ringers or Plasmalyte A) for intravenous fluid administration in the emergency department.

DETAILED DESCRIPTION:
The administration of intravenous fluids is ubiquitous in the care of the acutely ill. Commonly available isotonic crystalloid solutions contain a broad spectrum of electrolyte compositions including a range chloride concentrations. Recent studies have associated solutions with supraphysiologic chloride content with hyperchloremia, metabolic acidosis and renal vasoconstriction, acute kidney injury and renal replacement therapy, and increased mortality but no large, randomized-controlled trials have been conducted. SaLt-ED will be a large, cluster-randomized trial enrolling adults requiring intravenous isotonic crystalloid administration and hospital admission from the Vanderbilt University Emergency Department from January 1st 2016 until April 30 2017. The primary endpoint will be hospital-free days to day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Patient in the Vanderbilt Adult Emergency Department
2. Felt by treating clinician to require intravenous isotonic crystalloid
3. Felt by treating clinician to require inpatient hospital admission

Exclusion Criteria:

1. Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital-free days to day 28 | 28 days after enrollment
  The number of days alive and free of hospitalization in the first 28 days after study enrollment. Patients alive at the time of discharge will be presumed to be alive at 28 days. A patient who dies before hospital discharge will receive zero hospital-free days. A patient who remains in the hospital 28 days after enrollment will receive zero hospital-free days.

SECONDARY OUTCOMES:
Stage II or greater KIDNEY DISEASE IMPROVING GLOBAL OUTCOMES (KDIGO) Acute Kidney Injury | 30 days after enrollment censored at hospital discharge
  Proportion of patients with Stage II or greater acute kidney injury by KDIGO creatinine criteria (defined as rise in serum creatinine level of at least 2-fold, a serum creatinine level greater than or equal to 4.0 mg/dL with an acute increase of at least 0.5 mg/dL, or initiation of new renal replacement therapy).
Major adverse kidney event by hospital discharge or day 30 (MAKE30) | 30 days after enrollment
  At least one of: death, new renal replacement therapy, or persistent renal dysfunction at the time of hospital discharge (serum creatinine level ≥ 200% of baseline). Patients discharged prior to day 30 will be assumed not to develop this outcome between hospital discharge and day 30.
In-Hospital Mortality | 30 days or hospital discharge, whichever occurs first
  Death before hospital discharge
Hospital length of stay | Hospital length of stay assessed 90 days after enrollment
  Duration of hospitalization
ICU-free days to day 28 | 28 days
  Days alive and free of the intensive care unit in the first 28 days. Patients discharged prior to day 28 will be assumed to not have ICU days between discharge and day 28.
Ventilator-free days to day 28 | 28 days
  Days alive and free of mechanical ventilation in the first 28 days. Patients discharged prior to day 28 will be assumed to not have any ventilator days between discharge and day 28.
Vasopressor-free days | 28 days
  Days alive and free of vasopressor receipt in the first 28 days. Patients discharged prior to day 28 will be assumed to not have vasopressor days between discharge and day 28.
Receipt of new renal replacement therapy | 30 days after enrollment or hospital discharge, whichever occurs first
  Receipt of any form of renal replacement therapy in the first 30 days after enrollment in a patient who had not received renal replacement therapy prior to enrollment
Duration of new renal replacement therapy | 30 days after enrollment
  Duration of renal replacement therapy in the first 30 days after enrollment in a patient who had not received renal replacement therapy prior to enrollment
Peak creatinine | 28 days after enrollment or hospital discharge, whichever occurs first
  Highest creatinine in the 28 days after enrollment or hospital discharge, whichever occurs first
Change from baseline to peak creatinine | 28 days after enrollment or hospital discharge, whichever occurs first
  Change from baseline creatinine at enrollment to the highest creatinine before death or hospital discharge in the first 28 days
Incidence of metabolic acidosis and alkalosis | 30 days after enrollment or hospital discharge, whichever occurs first
  Incidence of metabolic acidosis and alkalosis in the first 30 days after enrollment as defined by bicarbonate values outside of the laboratory normal range.
Incidence of hyperchloremia and hypochloremia | 30 days after enrollment or hospital discharge, whichever occurs first
  Incidence of hyperchloremia and hypochloremia in the first 30 days after enrollment as defined by serum chloride values outside of the laboratory normal range.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Self, MD MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center Adult Emergency Department, Nashville, Tennessee, United States

REFERENCES:
- [Background] Finfer S, Liu B, Taylor C, Bellomo R, Billot L, Cook D, Du B, McArthur C, Myburgh J; SAFE TRIPS Investigators. Resuscitation fluid use in critically ill adults: an international cross-sectional study in 391 intensive care units. Crit Care. 2010;14(5):R185. doi: 10.1186/cc9293. Epub 2010 Oct 15. PMID 20950434
- [Background] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Background] Young P, Bailey M, Beasley R, Henderson S, Mackle D, McArthur C, McGuinness S, Mehrtens J, Myburgh J, Psirides A, Reddy S, Bellomo R; SPLIT Investigators; ANZICS CTG. Effect of a Buffered Crystalloid Solution vs Saline on Acute Kidney Injury Among Patients in the Intensive Care Unit: The SPLIT Randomized Clinical Trial. JAMA. 2015 Oct 27;314(16):1701-10. doi: 10.1001/jama.2015.12334. PMID 26444692
- [Derived] Self WH, Evans CS, Jenkins CA, Brown RM, Casey JD, Collins SP, Coston TD, Felbinger M, Flemmons LN, Hellervik SM, Lindsell CJ, Liu D, McCoin NS, Niswender KD, Slovis CM, Stollings JL, Wang L, Rice TW, Semler MW; Pragmatic Critical Care Research Group. Clinical Effects of Balanced Crystalloids vs Saline in Adults With Diabetic Ketoacidosis: A Subgroup Analysis of Cluster Randomized Clinical Trials. JAMA Netw Open. 2020 Nov 2;3(11):e2024596. doi: 10.1001/jamanetworkopen.2020.24596. PMID 33196806
- [Derived] Self WH, Semler MW, Wanderer JP, Wang L, Byrne DW, Collins SP, Slovis CM, Lindsell CJ, Ehrenfeld JM, Siew ED, Shaw AD, Bernard GR, Rice TW; SALT-ED Investigators. Balanced Crystalloids versus Saline in Noncritically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):819-828. doi: 10.1056/NEJMoa1711586. Epub 2018 Feb 27. PMID 29485926
- [Derived] Self WH, Semler MW, Wanderer JP, Ehrenfeld JM, Byrne DW, Wang L, Atchison L, Felbinger M, Jones ID, Russ S, Shaw AD, Bernard GR, Rice TW. Saline versus balanced crystalloids for intravenous fluid therapy in the emergency department: study protocol for a cluster-randomized, multiple-crossover trial. Trials. 2017 Apr 13;18(1):178. doi: 10.1186/s13063-017-1923-6. PMID 28407811